CLINICAL TRIAL: NCT02797132
Title: A Phase 3, 2-Part, Open-label Study to Evaluate the Safety and Pharmacokinetics of Lumacaftor/Ivacaftor Combination Therapy in Subjects Aged 2 Through 5 Years With Cystic Fibrosis, Homozygous for the F508del-CFTR Mutation
Brief Title: Safety and Pharmacokinetic Study of Lumacaftor/Ivacaftor in Subjects Aged 2 Through 5 Years With Cystic Fibrosis, Homozygous for F508del
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX15-809-115; 2016-001004-33 (EudraCT Number)
Record Dates: First submitted 2016-05-25; First posted 2016-06-13 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-09

CONDITIONS: Cystic Fibrosis
Keywords: CF
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor, ivacaftor drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lumacaftor/Ivacaftor (LUM/IVA) (Experimental): Part A (<14 kg): Participants weighing less than (<) 14 kilograms (kg) at screening received LUM 100 milligram (mg)/IVA 125 mg fixed-dose combination every 12 hours for 15 days in Part A.
  Part A (>=14 kg): Participants weighing greater than or equal to (>=) 14 kg at screening received LUM 150 mg/IVA 188 mg fixed-dose combination every 12 hours for 15 days in Part A.
  Part B (<14 kg): Participants weighing <14 kg at screening received LUM 100 mg/IVA 125 mg fixed-dose combination every 12 hours for 24 weeks in Part B.
  Part B (>=14 kg): Participants weighing >=14 kg at screening received LUM 150 mg/IVA 188 mg fixed-dose combination every 12 hours for 24 weeks in Part B.
  Interventions: Drug: LUM/IVA

INTERVENTIONS:
Drug: LUM/IVA
  Other Names: Orkambi; VX-809+VX-770

SUMMARY:
This is a Phase 3, 2-part (Part A and Part B), open-label, multicenter study evaluating the pharmacokinetics (PK), safety, tolerability, and pharmacodynamics (PD) of multiple doses of lumacaftor/ivacaftor (LUM/IVA) in subjects 2 through 5 years of age (inclusive) with cystic fibrosis (CF), homozygous for F508del. Subjects who participate in Part A may participate in Part B, if they meet the eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who weigh ≥8 kilogram (kg) without shoes and wearing light clothing at the Screening Visit
* Subjects with confirmed diagnosis of CF at the Screening Visit
* Subjects who are homozygous for the F508del-cystic fibrosis transmembrane conductance regulator (CFTR) mutation

Exclusion Criteria:

* Any clinically significant laboratory abnormalities at the Screening Visit that would interfere with the study assessments or pose an undue risk for the subject
* An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy (including antibiotics) for pulmonary disease within 28 days before Day 1
* A standard 12-lead ECG demonstrating QTc >450 millisecond (msec) at the Screening Visit.
* History of solid organ or hematological transplantation.
* Ongoing or prior participation in an investigational drug study (including studies investigating LUM and/or IVA) within 30 days of the Screening Visit.
* History of cataract/lens opacity or evidence of cataract/lens opacity determined to be clinically significant by a licensed ophthalmologist during the ophthalmologic examination at the Screening Visit

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (17):
  - Palo Alto, California
  - Aurora, Colorado
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - Buffalo, New York
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Houston, Texas
  - Norfolk, Virginia
  - Seattle, Washington
- Canada (3):
  - Vancouver, British Columbia
  - Toronto, Ontario
  - Montreal

REFERENCES:
- [Derived] McNamara JJ, McColley SA, Marigowda G, Liu F, Tian S, Owen CA, Stiles D, Li C, Waltz D, Wang LT, Sawicki GS. Safety, pharmacokinetics, and pharmacodynamics of lumacaftor and ivacaftor combination therapy in children aged 2-5 years with cystic fibrosis homozygous for F508del-CFTR: an open-label phase 3 study. Lancet Respir Med. 2019 Apr;7(4):325-335. doi: 10.1016/S2213-2600(18)30460-0. Epub 2019 Jan 24. PMID 30686767

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 2 parts, Part A and Part B. In Parts A and B, participants received doses of lumacaftor/ivacaftor (LUM/IVA) based on weight. Participants from Part A may have also participated in Part B.
Period: Part A (15 Days)
Arm/Group | Lumacaftor/Ivacaftor (LUM/IVA)
Started | 12
Part A (<14 kg Weight) | 4
Part A (>=14 kg Weight) | 8
Completed | 11
Not Completed | 1
Not completed — Adverse Event | 1
Period: Part B (24 Weeks)
Arm/Group | Lumacaftor/Ivacaftor (LUM/IVA)
Started | 60 (Participants from Part A may have participated in Part B.)
Part B (<14 kg Weight) | 19
Part B (>=14 kg Weight) | 41
Completed | 57
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: The Safety Set included all participants who received at least 1 dose of LUM/IVA in the respective study part.
Groups:
- Lumacaftor/Ivacaftor (LUM/IVA): Part A (<14 kg): Participants weighing <14 kg at screening received LUM 100 mg/IVA 125 mg fixed-dose combination every 12 hours for 15 days in Part A.
  Part A (>=14 kg): Participants weighing >=14 kg at screening received LUM 150 mg/IVA 188 mg fixed-dose combination every 12 hours for 15 days in Part A.
  Part B (<14 kg): Participants weighing <14 kg at screening received LUM 100 mg/IVA 125 mg fixed-dose combination every 12 hours for 24 weeks in Part B.
  Part B (>=14 kg): Participants weighing >=14 kg at screening received LUM 150 mg/IVA 188 mg fixed-dose combination every 12 hours for 24 weeks in Part B.
Arm/Group | Lumacaftor/Ivacaftor (LUM/IVA)
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: months] — Population: Data were planned to be reported separately for Part A and Part B of the study. Here "number analyzed" signifies participants who were evaluable for specified part of the study.
  months
    Part A (<14 kg Weight): number analyzed (Participants) | 4
    Part A (<14 kg Weight) | 27.0 (6.00)
    Part A (>=14 kg Weight): number analyzed (Participants) | 8
    Part A (>=14 kg Weight) | 48.0 (11.11)
    Part B (<14 kg Weight): number analyzed (Participants) | 19
    Part B (<14 kg Weight) | 31.6 (5.05)
    Part B (>=14 kg Weight): number analyzed (Participants) | 41
    Part B (>=14 kg Weight) | 49.9 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data were planned to be reported separately for Part A and Part B of the study. Here "number analyzed" signifies participants who were evaluable for specified part of the study.
  Participants
    Part A (<14 kg Weight): number analyzed (Participants) | 4
    Part A (<14 kg Weight): Female | 2
    Part A (<14 kg Weight): Male | 2
    Part A (>=14 kg Weight): number analyzed (Participants) | 8
    Part A (>=14 kg Weight): Female | 2
    Part A (>=14 kg Weight): Male | 6
    Part B (<14 kg Weight): number analyzed (Participants) | 19
    Part B (<14 kg Weight): Female | 9
    Part B (<14 kg Weight): Male | 10
    Part B (>=14 kg Weight): number analyzed (Participants) | 41
    Part B (>=14 kg Weight): Female | 20
    Part B (>=14 kg Weight): Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data were planned to be reported separately for Part A and Part B of the study. Here "number analyzed" signifies participants who were evaluable for specified part of the study.
  Participants
    Part A (<14 kg Weight): number analyzed (Participants) | 4
    Part A (<14 kg Weight): Hispanic or Latino | 0
    Part A (<14 kg Weight): Not Hispanic or Latino | 4
    Part A (<14 kg Weight): Unknown or Not Reported | 0
    Part A (>=14 kg Weight): number analyzed (Participants) | 8
    Part A (>=14 kg Weight): Hispanic or Latino | 0
    Part A (>=14 kg Weight): Not Hispanic or Latino | 8
    Part A (>=14 kg Weight): Unknown or Not Reported | 0
    Part B (<14 kg Weight): number analyzed (Participants) | 19
    Part B (<14 kg Weight): Hispanic or Latino | 1
    Part B (<14 kg Weight): Not Hispanic or Latino | 18
    Part B (<14 kg Weight): Unknown or Not Reported | 0
    Part B (>=14 kg Weight): number analyzed (Participants) | 41
    Part B (>=14 kg Weight): Hispanic or Latino | 2
    Part B (>=14 kg Weight): Not Hispanic or Latino | 39
    Part B (>=14 kg Weight): Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data were planned to be reported separately for Part A and Part B of the study. Here "number analyzed" signifies participants who were evaluable for specified part of the study.
  Participants
    Part A (<14 kg Weight): number analyzed (Participants) | 4
    Part A (<14 kg Weight): American Indian or Alaska Native | 0
    Part A (<14 kg Weight): Asian | 0
    Part A (<14 kg Weight): Native Hawaiian or Other Pacific Islander | 0
    Part A (<14 kg Weight): Black or African American | 0
    Part A (<14 kg Weight): White | 4
    Part A (<14 kg Weight): More than one race | 0
    Part A (<14 kg Weight): Unknown or Not Reported | 0
    Part A (>=14 kg Weight): number analyzed (Participants) | 8
    Part A (>=14 kg Weight): American Indian or Alaska Native | 0
    Part A (>=14 kg Weight): Asian | 0
    Part A (>=14 kg Weight): Native Hawaiian or Other Pacific Islander | 0
    Part A (>=14 kg Weight): Black or African American | 0
    Part A (>=14 kg Weight): White | 8
    Part A (>=14 kg Weight): More than one race | 0
    Part A (>=14 kg Weight): Unknown or Not Reported | 0
    Part B (<14 kg Weight): number analyzed (Participants) | 19
    Part B (<14 kg Weight): American Indian or Alaska Native | 0
    Part B (<14 kg Weight): Asian | 0
    Part B (<14 kg Weight): Native Hawaiian or Other Pacific Islander | 0
    Part B (<14 kg Weight): Black or African American | 0
    Part B (<14 kg Weight): White | 18
    Part B (<14 kg Weight): More than one race | 0
    Part B (<14 kg Weight): Unknown or Not Reported | 1
    Part B (>=14 kg Weight): number analyzed (Participants) | 41
    Part B (>=14 kg Weight): American Indian or Alaska Native | 0
    Part B (>=14 kg Weight): Asian | 0
    Part B (>=14 kg Weight): Native Hawaiian or Other Pacific Islander | 0
    Part B (>=14 kg Weight): Black or African American | 0
    Part B (>=14 kg Weight): White | 41
    Part B (>=14 kg Weight): More than one race | 0
    Part B (>=14 kg Weight): Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Pre-dose Concentration (Ctrough) of LUM and IVA
Time Frame: Day 15
Population: The pharmacokinetic (PK) set for Part A included all participants who received at least 1 dose of LUM/IVA in Part A.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Part A (<14 kg Weight): LUM 100 mg/IVA 125 mg: Participants weighing <14 kg at screening received LUM 100 mg/IVA 125 mg fixed-dose combination every 12 hours for 15 days in Part A.
- Part A (>=14 kg Weight): LUM 150 mg/IVA 188 mg: Participants weighing >=14 kg at screening received LUM 150 mg/IVA 188 mg fixed-dose combination every 12 hours for 15 days in Part A.
Arm/Group | Part A (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part A (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 4 | 7
nanogram per milliliter (ng/mL)
  LUM | 8710 (3590) | 12300 (5960)
  IVA | 94.0 (67.0) | 216 (185)

2. Primary Outcome: Part B: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 26
Population: The Safety Set included all participants who received at least 1 dose of LUM/IVA in Part B.
Measure: Count of Participants; unit: Participants
Groups:
- Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg: Participants weighing <14 kg at screening received LUM 100 mg/IVA 125 mg fixed-dose combination every 12 hours for 24 weeks in Part B.
- Part B (>=14 kg Weight): LUM 150 mg/IVA 188 mg: Participants weighing >=14 kg at screening received LUM 150 mg/IVA 188 mg fixed-dose combination every 12 hours for 24 weeks in Part B.
Arm/Group | Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part B (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 19 | 41
Participants
  AEs | 19 | 40
  SAEs | 2 | 2

3. Secondary Outcome: Part A: Pre-dose Concentration (Ctrough) of LUM and IVA Metabolites
Time Frame: Day 15
Population: The PK set for Part A included all participants who received at least 1 dose of LUM/IVA in Part A.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part A (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 4 | 7
ng/mL
  LUM Metabolite (M28 LUM) | 1310 (590) | 1370 (286)
  IVA Metabolite (M1 IVA) | 475 (384) | 1240 (1180)
  IVA Metabolite (M6 IVA) | 1510 (1130) | 3270 (2100)

4. Secondary Outcome: Part A: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Day 25
Population: The Safety Set included all participants who received at least 1 dose of LUM/IVA in Part A.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part A (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 4 | 8
Participants
  AEs | 4 | 6
  SAEs | 0 | 0

5. Secondary Outcome: Part B: Absolute Change From Baseline in Sweat Chloride at Week 24
Description: Sweat samples were collected using an approved collection device.
Time Frame: Baseline, Week 24
Population: The Full Analysis Set (FAS) included all enrolled participants in Part B who were exposed to any amount of LUM/IVA in Part B. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part B (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 18 | 31
millimole per liter (mmol/L) | -33.5 (14.5) | -30.7 (14.0)

6. Secondary Outcome: Part B: Absolute Change From Baseline in Body Mass Index (BMI) at Week 24
Description: BMI was defined as weight in kilograms (kg) divided by height in square meter (m^2).
Time Frame: Baseline, Week 24
Population: The FAS included all enrolled participants in Part B who were exposed to any amount of LUM/IVA in Part B. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Mean (Standard Deviation); unit: Kilogram per meter square (kg/m^2)
Arm/Group | Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part B (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 19 | 38
Kilogram per meter square (kg/m^2) | 0.22 (0.78) | 0.29 (0.75)

7. Secondary Outcome: Part B: Absolute Change From Baseline in Body Mass Index (BMI) For-Age Z-Score at Week 24
Description: BMI was defined as weight in kg divided by height in m^2. z-score is a statistical measure to describe whether a mean was above or below the standard. BMI, adjusted for age and sex, was analyzed as BMI-for-age z-score (BMI z-score).
Time Frame: Baseline, Week 24
Population: The FAS included all enrolled participants in Part B who were exposed to any amount of LUM/IVA in Part B. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part B (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 19 | 38
Z-score | 0.36 (0.67) | 0.26 (0.53)

8. Secondary Outcome: Part B: Absolute Change From Baseline in Weight at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part B (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 19 | 38
Kilogram (kg) | 1.4 (0.7) | 1.5 (1.0)

9. Secondary Outcome: Part B: Absolute Change From Baseline in Weight-for-age Z-Score at Week 24
Description: z-score is a statistical measure to describe whether a mean was above or below the standard. Weight, adjusted for age and sex, was analyzed as weight-for-age z-score (Weight z-score).
Time Frame: Baseline, Week 24
Population: The FAS included all enrolled subjects in Part B who were exposed to any amount of LUM/IVA in Part B. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part B (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 19 | 38
Z-score | 0.44 (0.52) | 0.17 (0.36)

10. Secondary Outcome: Part B: Absolute Change From Baseline in Stature (Height) at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part B (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 19 | 38
Centimeter (cm) | 4.1 (1.4) | 3.4 (1.0)

11. Secondary Outcome: Part B: Absolute Change From Baseline in Stature-for-Age Z-Score
Description: z-score is a statistical measure to describe whether a mean was above or below the standard. Stature (height), adjusted for age and sex, was analyzed as Stature-for-age z-score (Stature z-score).
Time Frame: Baseline, Week 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part B (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 19 | 38
Z-score | 0.19 (0.32) | 0.04 (0.19)

12. Secondary Outcome: Part B: Number of Pulmonary Exacerbations
Description: Pulmonary exacerbation was defined as new or changed treatment with oral, inhaled, or intravenous antibiotics and fulfillment of pre-specified protocol defined criteria.
Time Frame: Through Week 24
Population: as for outcome 6
Measure: Number; unit: pulmonary exacerbations
Arm/Group | Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part B (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 19 | 41
pulmonary exacerbations | 5 | 20

13. Secondary Outcome: Part B: Number of Participants With at Least One Pulmonary Exacerbation Pulmonary Exacerbation Through Week 24
Description: Pulmonary exacerbation was defined as new or changed treatment with oral, inhaled, or intravenous antibiotics and fulfillment of pre-specified protocol defined criteria. Time to event data was not collected and instead, number of participants with first event were collected and are reported. Time-to-first pulmonary exacerbation was planned to be estimated using Kaplan-Meier (KM) estimates. However, due to less than 50% of events, time-to-first event data was not estimated. Instead, number of participants with at least one pulmonary exacerbation event were collected and are reported.
Time Frame: Through Week 24
Population: The FAS included all enrolled participants in Part B who were exposed to any amount of LUM/IVA in Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part B (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 19 | 41
Participants | 3 | 15

14. Secondary Outcome: Part B: Number of Cystic Fibrosis (CF)-Related Hospitalizations
Time Frame: Through Week 24
Population: The FAS included all enrolled participants in Part B who were exposed to any amount of LUM/IVA in Part B.
Measure: Number; unit: hospitalizations
Arm/Group | Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part B (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 19 | 41
hospitalizations | 1 | 3

15. Secondary Outcome: Part B: Absolute Change From Baseline in Fecal Elastase-1 (FE-1) Levels at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: microgram per gram
Arm/Group | Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part B (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 12 | 23
microgram per gram | 38.4 (76.1) | 60.0 (94.0)

16. Secondary Outcome: Part B: Absolute Change From Baseline in Serum Levels of Immunoreactive Trypsinogen (IRT) Through Week 24
Time Frame: Baseline, Through Week 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg: Participants weighing less than 14 kg at screening received LUM 100 mg/IVA 125 mg fixed-dose combination every 12 hours for 24 weeks in Part B.
Arm/Group | Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part B (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 17 | 38
ng/mL | -262.1 (343.1) | -71.1 (120.5)

17. Secondary Outcome: Part B: Number of Participants With Microbiology Culture Status (Positive or Negative) at Week 24
Description: Following microbial tests were performed: Burkholderia, Methicillin Resistant Staphylococcus Aureus (MRSA), Methicillin Susceptible Staphylococcus Aureus (MSSA), Pseudomonas Aeruginosa Mucoid (P. Aeruginosa Mucoid), P. Aeruginosa Non-Mucoid, P. Aeruginosa Small Colony Variant and Stenotrophomonas Maltophilia.
Time Frame: Baseline and Week 24
Population: The FAS analysis set was used. Here "Number Analyzed" signifies those participants who were evaluated for this outcome at the specified time point..
Measure: Count of Participants; unit: Participants
Groups:
- Part B: LUM 100 mg/IVA 125 mg: Participants weighing less than <14 kg at screening received LUM 100 mg/IVA 125 mg fixed-dose combination every 12 hours for 24 weeks in Part B.
- Part B: LUM 150 mg/IVA 188 mg: Participants weighing >=14 kg at screening received LUM 150 mg/IVA 188 mg fixed-dose combination every 12 hours for 24 weeks in Part B.
Arm/Group | Part B: LUM 100 mg/IVA 125 mg | Part B: LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 19 | 41
Participants
  Baseline: Burkholderia: number analyzed (Participants) | 18 | 38
  Baseline: Burkholderia: Negative | 18 | 37
  Baseline: Burkholderia: Positive | 0 | 1
  Week 24: Burkholderia: number analyzed (Participants) | 19 | 36
  Week 24: Burkholderia: Negative | 19 | 36
  Week 24: Burkholderia: Positive | 0 | 0
  Baseline: MRSA: number analyzed (Participants) | 18 | 38
  Baseline: MRSA: Negative | 16 | 33
  Baseline: MRSA: Positive | 2 | 5
  Week 24:MRSA: number analyzed (Participants) | 19 | 36
  Week 24:MRSA: Negative | 17 | 35
  Week 24:MRSA: Positive | 2 | 1
  Baseline: MSSA: number analyzed (Participants) | 18 | 38
  Baseline: MSSA: Negative | 12 | 26
  Baseline: MSSA: Positive | 6 | 12
  Week 24: MSSA: number analyzed (Participants) | 19 | 36
  Week 24: MSSA: Negative | 13 | 26
  Week 24: MSSA: Positive | 6 | 10
  Baseline: P. Aeruginosa Mucoid: number analyzed (Participants) | 18 | 38
  Baseline: P. Aeruginosa Mucoid: Negative | 18 | 37
  Baseline: P. Aeruginosa Mucoid: Positive | 0 | 1
  Week 24: P. Aeruginosa Mucoid: number analyzed (Participants) | 19 | 36
  Week 24: P. Aeruginosa Mucoid: Negative | 19 | 35
  Week 24: P. Aeruginosa Mucoid: Positive | 0 | 1
  Baseline: P. Aeruginosa Non-Mucoid: number analyzed (Participants) | 18 | 38
  Baseline: P. Aeruginosa Non-Mucoid: Negative | 17 | 35
  Baseline: P. Aeruginosa Non-Mucoid: Positive | 1 | 3
  Week 24: P. Aeruginosa Non-Mucoid: number analyzed (Participants) | 19 | 36
  Week 24: P. Aeruginosa Non-Mucoid: Negative | 16 | 34
  Week 24: P. Aeruginosa Non-Mucoid: Positive | 3 | 2
  Baseline: P. Aeruginosa Small Colony Variant: number analyzed (Participants) | 18 | 38
  Baseline: P. Aeruginosa Small Colony Variant: Negative | 18 | 38
  Baseline: P. Aeruginosa Small Colony Variant: Positive | 0 | 0
  Week 24: P. Aeruginosa Small Colony Variant: number analyzed (Participants) | 19 | 36
  Week 24: P. Aeruginosa Small Colony Variant: Negative | 19 | 36
  Week 24: P. Aeruginosa Small Colony Variant: Positive | 0 | 0
  Baseline: Stenotrophomonas Maltophilia: number analyzed (Participants) | 18 | 38
  Baseline: Stenotrophomonas Maltophilia: Negative | 17 | 37
  Baseline: Stenotrophomonas Maltophilia: Positive | 1 | 1
  Week 24: Stenotrophomonas Maltophilia: number analyzed (Participants) | 19 | 36
  Week 24: Stenotrophomonas Maltophilia: Negative | 18 | 36
  Week 24: Stenotrophomonas Maltophilia: Positive | 1 | 0

18. Secondary Outcome: Part B: Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) at Week 24
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: Baseline, Week 24
Population: Analysis population: participants >=3 years of age with data available for Baseline and Week 24. Only participants from "Part B (>=14 Kg Weight)" arm met the eligibility criteria for the specified time point and were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part B (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 0 | 12
percentage of predicted FEV1 |  | 0.5 (11.6)

19. Secondary Outcome: Part B: Absolute Change in Sweat Chloride From Week 24 at Week 26
Description: Sweat samples were collected using an approved collection device.
Time Frame: Week 24, Week 26
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part B (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 17 | 31
mmol/L | 34.4 (14.9) | 32.2 (13.8)

20. Secondary Outcome: Part B: Acceptability/Palatability of LUM/IVA Granules Measured Using Hedonic Scale
Description: The acceptability and palatability of LUM/IVA granules was assessed by a visual analog scale that incorporates a 5 point facial hedonic scale (Liked it Very Much, Liked it a Little, Not sure, Disliked it a Little, Disliked it Very Much). The assessment was conducted in 2 steps: assessment of approved food/liquid (Evaluation 1), and assessment of approved food/liquid with LUM/IVA granules (Evaluation 2).
Time Frame: Day 1
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part B (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 18 | 38
Participants
  Evaluation 1: Liked it Very Much | 9 | 30
  Evaluation 1: Liked it a Little | 4 | 6
  Evaluation 1: Not sure | 3 | 1
  Evaluation 1: Disliked it a Little | 0 | 0
  Evaluation 1: Disliked it Very Much | 2 | 1
  Evaluation 2: Liked it Very Much | 4 | 6
  Evaluation 2: Liked it a Little | 2 | 5
  Evaluation 2: Not sure | 4 | 6
  Evaluation 2: Disliked it a Little | 3 | 6
  Evaluation 2: Disliked it Very Much | 5 | 15

21. Secondary Outcome: Part B: Absolute Change From Baseline in Lung Clearance Index (LCI) 2.5 at Week 24
Description: Lung clearance index (LCI) is a measure of ventilation inhomogeneity that is derived from a multiple breath washout test using Nitrogen (N2). LCI 2.5 represents the number of lung turnovers required to reduce the end tidal inert gas concentration to 1/40th of its starting value.
Time Frame: Baseline, Week 24
Population: The LCI Substudy Set included all participants who had signed informed consent (and assent, if applicable) to the optional LCI Substudy in Part B and enrolled and dosed in Part B. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part B (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 3 | 14
ratio | 0.27 (0.48) | -0.76 (1.19)

22. Secondary Outcome: Part B: Absolute Change From Baseline in Lung Clearance Index (LCI) 5.0 at Week 24
Description: LCI is a measure of ventilation inhomogeneity that is derived from a multiple breath washout test using Nitrogen (N2). LCI 5.0 represents the number of lung turnovers required to reduce the end tidal inert gas concentration to 1/20th of its starting value.
Time Frame: Baseline, Week 24
Population: The LCI Substudy Set included all subjects who had signed informed consent (and assent, if applicable) to the optional LCI Substudy in Part B and enrolled and dosed in Part B. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part B (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 3 | 14
ratio | 0.24 (0.40) | -0.12 (0.69)

23. Secondary Outcome: Part B: Pre-dose Concentration (Ctrough) of LUM and IVA and Its Metabolites
Time Frame: Week 24
Population: The PK set for Part B included all participants who received at least 1 dose of LUM/IVA in Part B. Here "Number Analyzed" signifies those participants who were evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B (<14 kg Weight): LUM 100 mg/IVA 125 mg | Part B (>=14 kg Weight): LUM 150 mg/IVA 188 mg
Number analyzed (Participants) | 19 | 41
ng/mL
  LUM: number analyzed (Participants) | 18 | 36
  LUM | 9060 (4060) | 9390 (4830)
  LUM Metabolite (M28 LUM): number analyzed (Participants) | 19 | 36
  LUM Metabolite (M28 LUM) | 1420 (846) | 1510 (752)
  IVA: number analyzed (Participants) | 18 | 35
  IVA | 108 (109) | 110 (108)
  IVA Metabolite (M1 IVA): number analyzed (Participants) | 18 | 36
  IVA Metabolite (M1 IVA) | 555 (560) | 521 (478)
  IVA Metabolite (M6 IVA): number analyzed (Participants) | 18 | 36
  IVA Metabolite (M6 IVA) | 2050 (1940) | 1900 (1430)

ADVERSE EVENTS:
Time Frame: Part A: Day 1 up to Day 25; Part B: Day 1 up to Week 26
Groups:
- Part A: LUM 100 mg/IVA 125 mg: Participants weighing <14 kg at screening received LUM 100 milligram (mg)/IVA 125 mg fixed-dose combination every 12 hours for 15 days in Part A.
- Part A: LUM 150 mg/IVA 188 mg: Participants weighing >= 14 kg at screening received LUM 150 mg/IVA 188 mg fixed-dose combination every 12 hours for 15 days in Part A.
- Part B: LUM 150 mg/IVA 188 mg: Participants weighing >=14 kg at screening received LUM 150 mg/IVA 188 mg fixed-dose combination every 12 hurs for 24 weeks in Part B.
Arm/Group | Part A: LUM 100 mg/IVA 125 mg | Part A: LUM 150 mg/IVA 188 mg | Part B: LUM 100 mg/IVA 125 mg | Part B: LUM 150 mg/IVA 188 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8 | 0/19 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8 | 2/19 | 2/41
Other Adverse Events (participants affected / at risk) | 4/4 | 6/8 | 19/19 | 40/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: LUM 100 mg/IVA 125 mg (N=4) | Part A: LUM 150 mg/IVA 188 mg (N=8) | Part B: LUM 100 mg/IVA 125 mg (N=19) | Part B: LUM 150 mg/IVA 188 mg (N=41)
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 0 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: LUM 100 mg/IVA 125 mg (N=4) | Part A: LUM 150 mg/IVA 188 mg (N=8) | Part B: LUM 100 mg/IVA 125 mg (N=19) | Part B: LUM 150 mg/IVA 188 mg (N=41)
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 7 | 10
Fatigue (General disorders) | 0 | 0 | 0 | 2
Chills (General disorders) | 0 | 0 | 1 | 1
Discomfort (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 0
Enuresis (Psychiatric disorders) | 0 | 0 | 0 | 1
Sleep terror (Psychiatric disorders) | 0 | 0 | 2 | 0
Tearfulness (Psychiatric disorders) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Radial head dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Respiratory rate increased (Investigations) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 3 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 4
Forced expiratory volume decreased (Investigations) | 0 | 0 | 0 | 2
Pseudomonas test positive (Investigations) | 0 | 0 | 3 | 2
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1
Burkholderia test positive (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 1
Pulmonary function test decreased (Investigations) | 0 | 0 | 0 | 1
Staphylococcus test positive (Investigations) | 0 | 0 | 0 | 1
Streptococcus test positive (Investigations) | 0 | 0 | 0 | 1
Bacterial test positive (Investigations) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 2 | 0
Blood iron decreased (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Enterovirus test positive (Investigations) | 0 | 0 | 1 | 0
Respirovirus test positive (Investigations) | 0 | 0 | 1 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 12 | 26
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 8 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 4
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 6 | 11
Constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Post-tussive vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Steatorrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Dyschezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 1 | 0 | 2
Lice infestation (Infections and infestations) | 0 | 1 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 3 | 7
Ear infection (Infections and infestations) | 0 | 0 | 3 | 4
Otitis media (Infections and infestations) | 0 | 0 | 0 | 4
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 3
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 2
Impetigo (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 2 | 1
Viral rash (Infections and infestations) | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 1
Candida nappy rash (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 1 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 2 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.

DOCUMENTS (2):
  • Study Protocol (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/32/NCT02797132/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT02797132/SAP_001.pdf